CLINICAL TRIAL: NCT06728956
Title: Assessing NHS ImplemeNTation of an onlinE Resilience Training Acceptance and Commitment Therapy (ACT) Programme to Prevent Job Loss in Multiple Sclerosis
Acronym: INTERACT-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NE24/164889
Record Dates: First submitted 2024-08-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main (Other): Participant outcomes will be measured at multiple time points (baseline, week 8 and month 6).
  assess for any change to outcome variables over time using repeated measures ANOVA, this provides only an overview of interventional impact and assumes homogenous change within the study group.
  Latent Growth Curve Modelling (LGCM) can be useful to identify patterns within subgroups of a population to understand who benefits from an intervention and why. Latent Growth Curve Modelling (LGCM) will be used to determine trajectories over time. Changes from baseline to week 8 and baseline to month 6 will be assessed.
  Interventions: Other: READY for MS UK digital programme

INTERVENTIONS:
Other: READY for MS UK digital programme — Online self-directed programme supported by HCPs

SUMMARY:
People with MS (PwMS) are at increased risk of leaving work earlier than expected. Psychological factors that affect PwMS may make it more difficult to manage staying in work. These can include psychological flexibility and self efficacy. Psychological flexibility is the ability to effectively manage unwanted inner experiences (e.g., thoughts, memories, bodily sensations) in the present. Self-efficacy is the self-belief that an individual has in their ability to succeed.

DETAILED DESCRIPTION:
Acceptance and Commitment Therapy (ACT) may help improve psychological flexibility and self-efficacy. Researchers and PwMS at Leeds have recently co-developed an online ACT-type programme called 'READY for MS'. This online programme may be helpful for PwMS who want to stay in work. READY for MS can be used on a computer or mobile device and does not need time off work traveling to see a psychologist. The aim is to understand the feasibility and effectiveness of training MS healthcare professionals to support delivery of the READY programme. Also to understand the long-term outcomes for both healthcare professionals and the PwMS they are supporting. What contexts contribute to effective delivery of the READY for MS programme will be explored. The aim is to test this READY for MS programme in various NHS settings to ensure that the programme is delivering the outcomes expected. This is a concept referred to as 'Intervention fidelity'. The key outcome that will be measured for PwMS is work instability (i.e. risk of job loss). Participants will be invited to complete online questionnaires. These will be completed at baseline, post-intervention and 6 month follow-up. The study team will invite a sub-set of participants to complete semi-structured interviews. The study team will use regular rapid qualitative analysis methods (lightning reports) to assess implementation.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving informed consent
* Age 18 years or above
* Currently in paid employment with an intention to remain in employment for at least 6 months
* Phase 2: A registered healthcare professional or allied health professional who works in direct contact with patients diagnosed with Multiple Sclerosis OR
* Phase 3: An individual with a clinical diagnosis of Multiple Sclerosis and reporting a WI score ≥11/22 (on MS-WIS)

Exclusion Criteria:

* Individuals lacking capacity to give informed consent
* Individuals intending to leave paid employment within the next 6 months
* Individuals who will not have access to a device used to access the internet (e.g.

laptop or smartphone) for the duration of study participation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Work Instability Scale (MS-WIS) | 6 months
  A 22-item psychometric validated self-report scale to measure work instability in multiple sclerosis. Work instability refers to any mismatch between job demands and an individual's functional (in)capacity and the extent to which this increases risk of job loss. Scores range from 0-22 and work instability is scored in bands of low risk (0-10), medium risk (11-16) and high risk (17-22).
Psychological Flexibility -Multi-dimensional Psychological Flexibility Inventory (MPFI) | 6 months
  a 60-item psychometric validated self-report scale to assess the key dimensions of flexibility and inflexibility from the Hexaflex model. For each sub-scale, items are scored 1-6 and then an average taken across the items of the sub-scale so that higher scores reflect higher levels of the dimension being assessed by each set of items. For the flexibility sub-scales, a higher score would indicate greater flexibility (better outcome) and for inflexibility sub-scales, higher scores indicate greater inflexibility (worse outcome).
Resilience Connor-Davidson Resilience Scale (CD-RISC 10) | 6 months
  A 10-item unidimensional psychometric validated self-report scale to measure resilience. Scores range 0-40 with a higher score indicating greater resilience (better outcome).
Self-efficacy -Unidimensional Self-efficacy scale for Multiple Sclerosis (USE-MS) | 6 months
  a 12-item psychometric validated self-report scale to measure self-efficacy in Multiple Sclerosis. Scores range 0-36 with a higher score indicating higher self-efficacy (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No